CLINICAL TRIAL: NCT05854966
Title: An Open Label, Pilot Phase II Study to Evaluate the Feasibility and Efficacy of CPI-613 Given With Metformin in Patients With Relapsed or Refractory Acute Myeloid Leukemia (AML)
Brief Title: CPI-613 Given With Metformin in Patients With Relapsed or Refractory Acute Myeloid Leukemia (AML)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI decided not to move forward with the study
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Cornerstone Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WFBCCC 22323; P30CA012197 (NIH)
Record Dates: First submitted 2023-05-02; First posted 2023-05-11 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Acute Myeloid Leukemia, in Relapse; Acute Myeloid Leukemia Refractory; Granulocytic Sarcoma
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Sarcoma, Myeloid | interventions — devimistat; Metformin; Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: This is a Phase II, Simon's two-stage study evaluating the feasibility and effectiveness of combination CPI-613 and metformin in relapsed or refractory acute myeloid leukemia. The first stage will consist of 9 evaluable patients. If the study continues to stage 2, a total of 17 evaluable patients will be enrolled.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment - CPI-613 with Metformin (Experimental): Induction therapy with CPI-613 and Metformin (ideally 2 hours prior to start of CPI-613 infusions on days 1-5) for two cycles of treatment.
  Maintenance therapy with CPI-613 and Metformin (ideally 2 hours prior to start of CPI-613 infusions on days 1-5) until progression, intolerable toxicity of withdrawal of consent.
  Interventions: Drug: CPI 613; Drug: Metformin; Biological: Blood draws; Procedure: Bone marrow biopsy

INTERVENTIONS:
Drug: CPI 613 — For INDUCTION therapy (14 day cycles): Devimistat (CPI-613) 2,500mg/m2, days 1-5, 14-day cycles for cycles 1 and 2 only.
  For MAINTENANCE therapy (21 day cycles): Devimistat (CPI-613) 2,500mg/m2, days 1-5, 21-day cycles until progression, intolerable toxicity or withdrawal of consent.
  Other Names: Devimistat
Drug: Metformin — For INDUCTION therapy (14 day cycles):
  Metformin 500 mg daily (taken with meals), days 1-2 for cycle 1 only. Metformin 500 mg twice daily (taken with meals), days 3-14 for cycle 1 only. Metformin 1,000 mg daily (taken with meals), days 1-2 for cycle 2 only. Metformin 1,000 mg twice daily (taken with meals) days 3-4 for cycle 2 only.
  For MAINTENANCE therapy (21 day cycles): Metformin 1,000 mg twice daily (taken with meals) days 1-21 until progression, intolerable toxicity or withdrawal of consent
  Other Names: Metformin pill
Biological: Blood draws — In the first induction cycle ONLY, extra blood will be withdrawn on day 1 before and after treatment with CPI-613 research purposes. Additional blood draws on days 2-5 to test blood before receiving CPI-613 to make sure participants are healthy enough to receive CPI-613.
Procedure: Bone marrow biopsy — After the second induction cycle participants will have a bone marrow biopsy. After this biopsy, participants will have other bone marrow biopsies every 3 months for the next year. After the first year, participants may have a bone marrow biopsy if the treating physician feels it is necessary.

SUMMARY:
The purpose of this research study is to find out what effects (the good and bad) the combination treatment of metformin and CPI-613 has in treating participants with acute myeloid leukemia or granulocytic sarcoma that has either returned after treatment or did not respond to treatment.

DETAILED DESCRIPTION:
Primary Objective: To establish the feasibility of delivering the combination of CPI-613 and metformin in patients with relapsed or refractory acute myeloid leukemia (AML).

Secondary Objectives: To determine the response rate of CPI-613 and metformin in relapsed or refractory AML defined as Complete remission (CR) + Complete remission with incomplete count recovery (CRi) + Morphologic Leukemia-Free State (MLFS).

* To determine the overall survival of patients with relapsed or refractory AML treated with CPI-613 and metformin.
* To determine the safety of CPI-613 and metformin in patients with relapsed or refractory acute myeloid leukemia (AML).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically documented relapsed and/or refractory Acute Myeloid Leukemia or granulocytic sarcoma.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 3.
* Must be ≥ 18 years of age.
* Persons of child-bearing potential (i.e., women who are pre-menopausal or not surgically sterile) must use accepted contraceptive methods (abstinence, intrauterine device [IUD], oral contraceptive or double barrier device), and must have a negative serum or urine pregnancy test within 1 week prior to treatment initiation.
* Persons who are having sexual relationships in which their partner may become pregnant must practice effective contraceptive methods during the study treatment and for 60 days after the last dose of study treatment, unless documentation of infertility exists.
* Mentally competent, ability to understand and willingness to sign the informed consent form.
* Patients with persisting, non-hematologic, non-infectious toxicities from prior treatment must be ≤ Grade 2 and must be documented as such.
* Laboratory values ≤ 2 weeks prior to the start of study treatment must be the following:
* Aspartate aminotransferase [AST/SGOT] ≤ 5x upper normal limit [UNL],
* Alanine aminotransferase [ALT/SGPT] ≤ 5x UNL
* Bilirubin ≤ 3x UNL
* Albumin ≥ 2.0 g/dL or ≥ 20 g/L
* Serum creatinine ≤ 2.0 mg/dL
* Presence of central venous catheter or willing to have central venous access placed.

Exclusion Criteria:

* Patients with active central nervous system (CNS) or epidural tumor.
* Pregnant persons, or persons of child-bearing potential not using reliable means of contraception (because the teratogenic potential of CPI-613 is unknown).
* Breastfeeding individuals because the potential of excretion of CPI-613 into breast milk. (Note: Breastfeeding individuals are excluded because the effects of CPI-613 on a nursing child are unknown).
* Any condition or abnormality which may, in the opinion of the investigator, compromise the safety of patient.
* Unwilling or unable to follow protocol requirements.
* Patients receiving any other standard or investigational treatment for their cancer, or any other investigational agent for any indication within the past 1 week prior to initiation of CPI-613 treatment with the following exceptions:
* The use of Hydrea or any targeted oral agent is allowed up to the day before initiation of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Number of Participants to Receive at Least One Cycle of Maintenance Therapy - Feasibility | After the completion of cycle 1 of maintenance therapy (maintenance cycle is 21 days)
  Feasibility is defined as the ability to deliver at least 1 cycle of maintenance therapy in 50% or more of patients who complete induction therapy.

SECONDARY OUTCOMES:
Response Rate - Efficacy (Acute Myeloid Leukemia European LeukemiaNet 2022) | After the completion of cycle 2 (each cycle is 14 days), then every three months up to 12 months
  Efficacy will be assessed in the first 9 evaluable participants using a Simon's two-stage design to examine efficacy in terms of response where response is defined as:
  * Complete remission (CR) (Bone marrow blasts, 5%; absence of circulating blasts; absence of extramedullary disease; ANC ≤ 1.0 × 109/L (1,000/μL); plate) or
  * Complete remission with incomplete count recovery (CRi) (All CR criteria except for residual neutropenia < 1.0 × 109/L (1,000/μL) or thrombocytopenia < 100 × 109/L (100,000/μL) or
  * Morphologically leukemia free state (MLFS) (Bone marrow blasts < 5%; absence of circulating blasts; absence of extramedullary disease; no hematologic recovery required).
Overall Survival | Every 3 months after last dose of study treatment, up to 2 years
  Overall survival is calculated in days from date of study treatment initiation to date of death due to any cause. Patients last known to be alive are censored at date of last contact.
Number of Reported Adverse Events - Safety | Up to 30 days after last dose of study treatment
  Safety will be evaluated by describing the nature and frequency of adverse events as defined by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Bayard Powell, MD, Principal Investigator — Wake Forest Baptist Comprehensive Cancer Center

IPD SHARING:
Plan to Share IPD: No